CLINICAL TRIAL: NCT00571922
Title: A Placebo-controlled, Double Blind, Randomized Trial of Acamprosate for the Treatment of Methamphetamine Dependence
Brief Title: A Clinical Trial of Acamprosate for Treatment of Methamphetamine Addiction
Acronym: AcampMet
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: Forest Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 06-632
Record Dates: First submitted 2007-12-10; First posted 2007-12-12 (Estimated); Results first posted 2016-04-06 (Estimated); Last update posted 2017-03-24 (Actual); Status verified 2017-03

CONDITIONS: Methamphetamine Dependence, Treatment Seeking
Keywords: methamphetamine, crystal, treatment
MeSH Terms: interventions — Acamprosate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Acamprosate (Active Comparator)
  Interventions: Drug: Acamprosate
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Acamprosate — 2 gr/day (333 mg, TID)
  Other Names: Campral
  Arms: Acamprosate
Drug: placebo — matching placebo
  Arms: Placebo

SUMMARY:
This clinical trial will compare 10 week treatment with acamprosate (2 gr/day) versus placebo, combined with weekly abstinence oriented individual counseling, in methamphetamine dependent patients, 72 subjects will be enrolled, with an interim analysis scheduled after 36 enrolled. Primary outcome is methamphetamine absitience over the 10 week treatment period, and the last 2 weeks of treatment. Abstinence is defined on a weekly basis as no urine positive of methamphetamine (or amphetamine) and self-report of not use for the 7 day period. Secondary measures include treatment retention, drug craving, mood, and safety.

ELIGIBILITY:
Inclusion Criteria:

* Methamphetamine dependence
* Treatment seeking
* Urine sample (+) for methamphetamine

Exclusion Criteria:

* Pregnancy
* Dependence on other drugs (except nicotine)
* DSM-IV axis I disorder unrelated to drug abuse
* Serious medical condition in clinicians opinion.
* AIDs
* Untreated syphilis
* Allergy to acamprosate
* Methadone, or other ORP, maintenance

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2007-07; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Malcolm Reid, PhD, Principal Investigator — NYU Langone Health
Locations (1):
- VA New York Harbor Healthcare System, MHAD clinic, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Acamprosate | Placebo
Started | 36 | 36
Completed | 0 | 0
Not Completed | 36 | 36
Not completed — Completion unknown | 36 | 36

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Acamprosate | Placebo | Total
Number analyzed (Participants) | 36 | 36 | 72
Age, Categorical [Count of Participants; unit: Participants] — PI passed away, and there is no access to data. Although the total number of subjects enrolled is known, information regarding baseline characteristics is unavailable.
  Participants
    <=18 years | NA — PI passed away, and there is no access to data. Although the total number of subjects enrolled is known, information regarding baseline characteristics is unavailable. | NA — PI passed away, and there is no access to data. Although the total number of subjects enrolled is known, information regarding baseline characteristics is unavailable. | NA — Total not calculated because data are not available (NA) in one or more arms.
    Between 18 and 65 years | NA — PI passed away, and there is no access to data. Although the total number of subjects enrolled is known, information regarding baseline characteristics is unavailable. | NA — PI passed away, and there is no access to data. Although the total number of subjects enrolled is known, information regarding baseline characteristics is unavailable. | NA — Total not calculated because data are not available (NA) in one or more arms.
    >=65 years | NA — PI passed away, and there is no access to data. Although the total number of subjects enrolled is known, information regarding baseline characteristics is unavailable. | NA — PI passed away, and there is no access to data. Although the total number of subjects enrolled is known, information regarding baseline characteristics is unavailable. | NA — Total not calculated because data are not available (NA) in one or more arms.
Sex: Female, Male [Count of Participants; unit: Participants] — PI passed away, and there is no access to data. Although the total number of subjects enrolled is known, information regarding baseline characteristics is unavailable.
  Participants
    Female | NA — PI passed away, and there is no access to data. Although the total number of subjects enrolled is known, information regarding baseline characteristics is unavailable. | NA — PI passed away, and there is no access to data. Although the total number of subjects enrolled is known, information regarding baseline characteristics is unavailable. | NA — Total not calculated because data are not available (NA) in one or more arms.
    Male | NA — PI passed away, and there is no access to data. Although the total number of subjects enrolled is known, information regarding baseline characteristics is unavailable. | NA — PI passed away, and there is no access to data. Although the total number of subjects enrolled is known, information regarding baseline characteristics is unavailable. | NA — Total not calculated because data are not available (NA) in one or more arms.

OUTCOME MEASURES:

1. Primary Outcome: Methamphetamine Abstinence
Time Frame: 7 day
Population: PI passed away, data is unavailable.
Arm/Group | Acamprosate | Placebo
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Craving
Time Frame: 7 day
Population: PI passed away, data is unavailable
Arm/Group | Acamprosate | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: PI passed away, and there is no access to data. Information regarding adverse and serious adverse events is unavailable.
Arm/Group | Acamprosate | Placebo
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Sadly, the PI of this study passed away on 4/20/2010. Data was not analyzed and is unavailable.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes